CLINICAL TRIAL: NCT02179528
Title: Phase 2 Study of Small Doses of Etoposide as Maintenance Treatment in Small Cell Lung Cancer
Brief Title: Study of Small Doses of Etoposide as Maintenance Treatment in Small Cell Lung Cancer(SCLC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jie Wang, Chief of thoracic cancer department, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJCHDTC001
Record Dates: First submitted 2014-06-24; First posted 2014-07-02 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-06

CONDITIONS: Small Cell Lung Cancer Extensive Stage
MeSH Terms: interventions — Etoposide

ARMS (2):
- etoposide,maintenance therapy (Active Comparator): etoposide,25mg qd d1-20，repeat every 28 days
  Interventions: Drug: Etoposide
- blank control (No Intervention): blank control

INTERVENTIONS:
Drug: Etoposide
  Arms: etoposide,maintenance therapy

SUMMARY:
Patients with extensive-stage small cell lung cancer receive six cycles of chemotherapy(etoposide plus platinum) as first-line treatment,who achieve Complete Response(CR)/Partial Response(PR) will accept small doses of etoposide as maintenance treatment. The objective of this study is to evaluate the progression free survival,overall survival,objective response rate,disease control rate and safety of etoposide as maintenance therapy. Based on previous studies on maintenance therapy in small cell lung cancer,the hypothesis of this study is maintenance therapy using etoposide may improve progression free survival,overall survival for selected patients. The investigators will use the peripheral blood to assess circulating tumor cell and cell-free DNA,which may help us to screen a subgroup of patients with better response to etoposide maintenance therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of small cell lung cancer
* Extensive stage according to American Veteran Staging System
* At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST )1.1
* Eastern Cooperative Oncology Group (ECOG) scores for performance status of 0 to 2
* Age≥18 years
* Adequate organ function
* Consent form according with Guideline for Good Clinical Practice of the International Conference on Harmonisation (ICH-GCP)guidelines
* The expected survival≥2 months

Exclusion Criteria:

* Pathological diagnosis of mixed small cell lung cancer
* Limited stage according to American Veteran Staging System
* Other preexisting or existing malignant tumors,not including non-melanoma skin cancer with effective treatment,cervical cancer in situ or tumor response has been 3 years which is considered cured by the investigator
* Known pre-existing interstitial lung disease
* Pre-existing or uncontrolled gastrointestinal disease which may affect drug absorption or worsen existing disease believed by the investigator
* Any other medical history or coexisting disease that may affect compliance of patients or the assessment of safety and effectiveness of the drug believed by the investigator
* Pregnant or lactating women
* Active phase of hepatitis B virus infection,Active phase of hepatitis C virus infection or known HIV carriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Time to Disease Progression | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, doctor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhang C, Duan J, He Z, Yang L, Yang S, Zhang Z, Liu Y, Wan R, Lin L, Wu X, Wang W, Wang Q, Wang J. The benefits of etoposide capsules as maintenance therapy for patients with extensive-stage small cell lung cancer: a prospective two-stage, two-center study. J Thorac Dis. 2021 Jan;13(1):343-352. doi: 10.21037/jtd-21-106. PMID 33569214